CLINICAL TRIAL: NCT05979571
Title: Development of Educational Intervention Through Technological Platform to Support Exclusive Breastfeeding up to Six Months Pilot Study
Brief Title: Developing and Testing an Educational Intervention Through Technological Platform to Support Exclusive Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pacifica Salud Hospital (Network)
Collaborators: Sistema Nacional de Investigación Senacyt Panamá (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2880
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Breastfeeding, Exclusive
Keywords: breastfeeding, mobile health, perinatal care, primary care
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Other: Mobile health app

INTERVENTIONS:
Other: Mobile health app — Breastfeeding knowledge and promotion information will be delivered through the AmiBreastfeed app platform

SUMMARY:
Although breastfeeding provides the infant with all the nutrients necessary for its development, it has been observed that in Panama there are low rates of Exclusive Breastfeeding. Educational interventions, that support exclusive breastfeeding, which begin before delivery and continue to the postnatal period, have been shown to be effective.

The main objective of the study is the development and testing of an educational intervention through web based platform, to support exclusive breastfeeding up to 6 months. This educational intervention will provide guidance with the help of an audiovisual format, with information and breastfeeding techniques, which mothers can reproduce as many times as necessary.

The main objective of the study is the development and testing of an educational intervention through AmiHealth, to support exclusive breastfeeding up to 6 months.

A pilot study will be conducted on a non-random convenience sample.

DETAILED DESCRIPTION:
The team leveraged a user-centered design (UCD) approach to design and develop the initial version of the breastfeeding app. An agile development methodology for content and technology development which integrates feedback from all key stakeholders in the development process to refine the app over time, including the content and app.In parallel with the app design, the educational content for the intervention was developed with experts in the field.

The contents that will be develop for the breastfeeding module, Data operating system will be used for data management and analytical and projection tools.

ELIGIBILITY:
Inclusion Criteria:

1. First pregnancy
2. Third trimester

Exclusion Criteria:

* twin pregnancies fetal defects or newborns with malformations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Mobile application rating scale (MARS) | two weeks
  The quality of the apps will be asses using MARS. This methodology includes 23 evaluation criteria, clustered within 5 domains: (1) "Engagement," which assesses the entertainment, customization, and interactivity of the app (feedback, reminders, and notifications); (2) "Functionality," which examines the functionality of the app, ease of use, transition between screens, and intuitive design; (3) "Esthetics," which assesses graphic design, visual appeal, and stylistic consistency; (4) "Information," which evaluates the quality of the content (text, measures, and references), determined by the credibility of the source; and (5) "Subjective quality," which determines whether the app could be recommended to people who might benefit from it, if they would be prepared to pay for it, how many times it would be used, and what overall star rating it would be given. Each evaluation criterion was rated from 1 to 5 (1=Inadequate, 2=Poor, 3=Acceptable, 4=Good, 5=Excellent)

CONTACTS AND LOCATIONS:
Overall Officials: Tania T Herrera, MD, Principal Investigator — Pacifica Salud Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meedya S, Fernandez R, Fahy K. Effect of educational and support interventions on long-term breastfeeding rates in primiparous women: a systematic review and meta-analysis. JBI Database System Rev Implement Rep. 2017 Sep;15(9):2307-2332. doi: 10.11124/JBISRIR-2016-002955. PMID 28902698
- [Result] Spatz DL, Davanzo R, Muller JA, Powell R, Rigourd V, Yates A, Geddes DT, van Goudoever JB, Bode L. Promoting and Protecting Human Milk and Breastfeeding in a COVID-19 World. Front Pediatr. 2021 Feb 3;8:633700. doi: 10.3389/fped.2020.633700. eCollection 2020. PMID 33614547
- [Result] Vu Hoang D, Cashin J, Gribble K, Marinelli K, Mathisen R. Misalignment of global COVID-19 breastfeeding and newborn care guidelines with World Health Organization recommendations. BMJ Nutr Prev Health. 2020 Dec 22;3(2):339-350. doi: 10.1136/bmjnph-2020-000184. eCollection 2020 Dec. PMID 33521544
- [Result] Huang MZ, Kuo SC, Avery MD, Chen W, Lin KC, Gau ML. Evaluating effects of a prenatal web-based breastfeeding education programme in Taiwan. J Clin Nurs. 2007 Aug;16(8):1571-9. doi: 10.1111/j.1365-2702.2006.01843.x. PMID 17655546
- [Result] Alberdi G, O'Sullivan EJ, Scully H, Kelly N, Kincaid R, Murtagh R, Murray S, McGuinness D, Clive A, Brosnan M, Sheehy L, Dunn E, McAuliffe FM. A feasibility study of a multidimensional breastfeeding-support intervention in Ireland. Midwifery. 2018 Mar;58:86-92. doi: 10.1016/j.midw.2017.12.018. Epub 2017 Dec 24. PMID 29324318
- See also: Unicef Breastfeeding Information — https://www.unicef.org/media/48046/file/UNICEF_Breastfeeding_A_Mothers_Gift_for_Every_Child.pdf
- See also: Sexual and Reproductive Health survey 2014-2015 — https://panama.unfpa.org/sites/default/files/pub-pdf/ENASSER-2014-2015-WEB.pdf